CLINICAL TRIAL: NCT07352020
Title: Evaluation of Platelet Rich Plasma in Reducing Sternal Wound Complications in CABG Surgery With Median Sternotomy
Brief Title: Use of Platelet-Rich Plasma to Reduce Sternal Wound Complications After CABG With Median Sternotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Sangeen khan Wazir, Registrar, Cardiac Surgery, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-4/AS&RB-M/SZABMU/2022-; F.1-1/2015/ERB/SZAMU/932 (Other: Shaheed Zulfiqar Ali Bhutto Medical University)
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Surgical Site Infection (SSI); Mediastinitis; Delayed Wound Healing
Keywords: Sternal wound infection; Superficial sternal wound infection; Deep sternal wound infection; Surgical site infection; Delayed wound healing; Median sternotomy; Cardiac surgery; Postoperative wound complications; Hospital length of stay; Cost analysis; Platelet rich plasma; coronary artery bypass grafting; wound healing; CABG; readmission rate
MeSH Terms: conditions — Surgical Wound Infection; Mediastinitis

STUDY DESIGN:
Intervention Model Description: This interventional study uses a parallel group design. Participants undergoing median sternotomy are randomized to one of two study arms: standard sternal wound closure or autologous platelet-rich plasma (PRP) applied before standard sternal wound closure. Each participant receives only the assigned intervention. Participants and outcome assessors are blinded to group assignment, while surgeons performing the procedure are aware of the intervention. Postoperative outcomes, including primary outcomes as superficial & deep sternal wound infections, delayed wound healing and rate of readmissions. Secondary outcome as cost (pre-specified secondary outcome) and other observed outcomes such as length of ICU stay, RCC used more than 4 units, platelets used more than 4 units are compared between groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to group assignment. Surgeons performing the procedure and the study investigator are aware of the intervention to ensure proper delivery of PRP and adherence to the study protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Sternal Wound Closure (Active Comparator): Conventional sternal wound closure is performed without platelet-rich plasma. Participants and outcome assessors are blinded to group assignment; surgeons are aware of the intervention. Postoperative outcomes including superficial and deep sternal wound infections, delayed wound healing, cost (pre-specified secondary outcome), rate of admissions, and other observed outcomes such as length of hospital stay and more than 4 units of RCC & platelets were assessed.
  Interventions: Procedure: Standard Sternal Wound Closure
- PRP with Standard Sternal Wound Closure (Experimental): Autologous platelet-rich plasma (6 ml) is applied to the sternal wound before closure. Participants and outcome assessors are blinded to group assignment; surgeons are aware of the intervention. Postoperative outcomes including superficial and deep sternal wound infections, delayed wound healing, cost (pre-specified secondary outcome), rate of admissions, and other observed outcomes such as length of hospital stay and more than 4 units of RCC & platelets were assessed.
  Interventions: Procedure: Autologous Platelet-Rich Plasma (PRP) Application

INTERVENTIONS:
Procedure: Autologous Platelet-Rich Plasma (PRP) Application — Autologous platelet-rich plasma (PRP) is prepared from the patient's own blood and applied directly to the sternal wound before standard surgical closure during cardiac surgery. The PRP contains concentrated platelets and growth factors intended to enhance wound healing and reduce infection risk. Patients in this arm receive standard sternal closure after PRP application. The procedure is performed in the operating room after sternotomy and prior to wound closure. The application is performed by the surgeon following standardized protocol to ensure consistent delivery across all participants. This intervention differs from standard closure alone and is intended to improve postoperative wound outcomes.
  Arms: PRP with Standard Sternal Wound Closure
Procedure: Standard Sternal Wound Closure — Patients in this arm receive the standard surgical closure of the sternal wound following median sternotomy for cardiac surgery. No experimental or additional biologic products are applied. The procedure is performed according to routine surgical protocols used at the study site. This arm serves as the control group, allowing comparison of outcomes such as wound healing, infection rates, ICU stay, hospitalization cost and more than 4 units of RCC & platelets were assessed with the experimental arm receiving platelet-rich plasma (PRP) application.
  Arms: Standard Sternal Wound Closure

SUMMARY:
The goal of this clinical trial is to learn whether applying autologous platelet-rich plasma (PRP) to the sternal wound during heart surgery improves wound healing and reduces complications after surgery. The study also aims to evaluate whether PRP can reduce hospital-related outcomes and costs.

The main questions this study aims to answer are:

Does the use of PRP reduce superficial & deep sternal wound infections and rate of readmissions?

Does PRP improve wound healing after heart surgery?

Does PRP reduce the cost of hospitalization and length of ICU stay.

Does PRP reduce the requirement of red cell concentrate (RCC) and platelets to less than 4 units each

Researchers will compare PRP applied to the sternal wound before closure with standard sternal wound closure alone to determine whether PRP provides additional benefit beyond standard surgical care.

Participants were randomly assigned to one of two groups.

Participants will:

Receive standard sternal wound closure or PRP applied to the sternal wound followed by standard closure

Be monitored for wound infections and healing outcomes after surgery

Have hospital cost, RCC & platelet units used, ICU stay, and readmission data recorded during the postoperative period

Patients and outcome assessors were blinded to the treatment assignment. Surgeons were aware of the intervention due to the nature of the procedure.

This study aims to determine whether adding PRP to standard sternal closure can improve recovery and reduce complications following cardiac surgery.

DETAILED DESCRIPTION:
Official Title:

Evaluation of Platelet Rich Plasma in Reducing Sternal Wound Complications in CABG Surgery With Median Sternotomy.

Study Background:

Median sternotomy is the standard approach for most cardiac surgeries, providing low failure rates and good long-term outcomes. However, complications such as wound infection, sternal dehiscence, and delayed healing, although uncommon, can lead to serious morbidity, longer hospital stays, and increased costs. Risk factors include obesity, diabetes, smoking, steroid use, osteoporosis, chronic lung disease, and mobilization of the internal mammary arteries. Platelet-rich plasma (PRP), which contains concentrated platelets and growth factors, has shown promise in promoting tissue healing, reducing infections, and supporting bone regeneration. PRP is used in various surgical fields but is not yet routine in cardiac surgery. Early studies suggest that applying PRP during sternotomy may reduce postoperative sternal wound complications and the need for reoperation.

Rationale:

Postoperative complications are a significant cause of morbidity in patients undergoing cardiac surgery. Platelet-rich plasma has been proposed in clinical studies as an adjunctive therapy to reduce the incidence of complications in patients undergoing cardiac procedures via median sternotomy. The purpose of this study is to evaluate the potential benefit of platelet-rich plasma, in addition to standard care, in patients undergoing on-pump coronary artery bypass graft surgery.

Brief Summary:

This study will test whether applying a patient's own platelet-rich plasma (PRP) to the breastbone area during heart surgery can help wounds heal better after coronary artery bypass surgery. Ninety-eight patients will be randomly assigned to standard closure or closure with PRP, and the study will track healing, infections, hospital stay, blood transfusions, and related costs for 30 days. The goal is to see if PRP can reduce complications and improve recovery after surgery.

Detailed description:

The effect of autologous platelet-rich plasma (PRP) in this randomized controlled trial will be studied on postoperative sternal wound complications in patients undergoing on-pump coronary artery bypass graft surgery via median sternotomy. The study will enroll 98 patients aged 45 to 72 years who provide informed consent. Participants will be recruited consecutively and randomly assigned to one of two groups. All patients will undergo standard sternal closure using a midline sternotomy with a sternal saw blade, closure of the sternum with simple interrupted or figure-of-eight stainless steel wires, and layered wound closure with absorbable sutures, followed by standard dressing with Steri-Strips, gauze, and paper tape. The intervention group will additionally receive 6 mL of autologous PRP applied to the sternum and surrounding soft tissue during sternal closure. Both participants and outcome assessors will be blinded to group assignment, while surgeons performing the procedures will be aware of the intervention. The study aims to determine whether the addition of PRP to standard care reduces the frequency of sternal wound complications compared with standard sternal closure alone. All participants will provide written informed consent, and their confidentiality will be maintained. Standard care will not be altered for study purposes.

Study Design:

This is an interventional, randomized, parallel-assignment trial with double blinding (participants and outcome assessors), while the surgeons performing the procedures will be aware of the intervention. The primary purpose of the study is treatment. Participants will be randomly assigned to standard sternal closure or sternal closure with PRP.

Eligibility Criteria:

Consenting patients from 45 to 72 years of age, undergoing on pump CABG surgery with median sternotomy.

Patients will be excluded if they have a body mass index less than 18.5 or greater than 24.9, have undergone bilateral harvesting of the internal mammary artery, are receiving steroid therapy, have a known diagnosis of diabetes mellitus, are active smokers, have osteoporosis or chronic lung disease, have a cardiopulmonary bypass time exceeding 72.5 minutes, are unable to have platelet-rich plasma prepared, or are not eligible for blood bank donation.

Sample size

The sample size was calculated based on the primary outcome of sternal wound complications within 30 days post-surgery. Using the WHO sample size calculator with the following assumptions:

Level of significance (α) = 5% Power (1-β) = 80% Proportion of sternal wound complications in PRP group (P1) = 18% Proportion of sternal wound complications in control group (P2) = 44% The required sample size is 49 patients per group, for a total of 98 patients. This calculation ensures adequate statistical power to detect a clinically meaningful reduction in postoperative sternal wound complications between the PRP and control groups.

Outcome Measures:

Primary Outcome:

Frequency of sternal wound complications (delayed healing, superficial and deep infections, readmission including mediastinitis) within 30 days.

Secondary Outcome:

Overall cost burden (additional medications, additional antibiotics, additional laboratory tests, additional wound care, additional surgical procedure) during the 30-day postoperative period.

Other Outcomes:

ICU stay (days), red cell transfusions >4 units, platelet transfusions >4 units.

OPERATIONAL DEFINITIONS

DSWI:

DSWI diagnosis will be made, based on the guidelines of the CDC, in patients who developed one or more of the following: positive culture of mediastinal tissue or fluid; clinical evidence of mediastinitis during sternal reoperation; or chest pain, sternal instability, purulent discharge from the mediastinum associated with a positive blood culture. DSWI presenting in the first 30 days after operation will be included in the study.

SWI:

All the infections will be considered positive that will involve skin and subcutaneous tissue within the first 30 postoperative days, not reaching the sternum, requiring local surgical intervention with regular wound care, accompanied by antibiotic therapy and/or Vacuum Assisted Closure (VAC) therapy.

Delayed Healing:

Healing is a complex biochemical process of tissue repair after it has been damaged. It has three stages which are inflammation, proliferation and remodelling. Delay in the specific time period or in the biochemical process is called delayed healing. Skin, subcutaneous tissue or sternum which is unable to heal within two weeks of surgery will be considered delayed wound healing.

Readmission:

It is defined as any hospital readmission within 30 days of discharge related to the index surgery.

ICU stay:

Stay that refers to the duration, in days, spent in the intensive care unit, within 30 days postoperatively.

Blood transfusion:

It is defined as the requirement of more than 4 units of packed red blood cells (PRBC) or platelets within 30 days postoperatively.

Data Collection Procedure:

The study protocol will be submitted for approval to the hospital ethics committee and Advance Research Committee, and written informed consent will be obtained from all participants. Eligible patients will be enrolled from the Cardiac Center and recruited consecutively, then randomly assigned to either the control group (standard sternal closure) or the intervention group (standard closure plus 6 mL of autologous PRP applied to the sternum and soft tissue). Standard perioperative care, including antibiotic prophylaxis, glycemic management, and general anesthesia, will be applied to all patients. Surgery will be performed via midline sternotomy, with cardiopulmonary bypass according to local guidelines, and heparinization maintained to an activated clotting time ≥480 s. Bone wax will be avoided to prevent interference with PRP. Following closure with stainless steel wires and layered sutures, standard dressings will be applied. Participants and outcome assessors will be blinded to group assignment, while surgeons will be aware of the intervention. All data will be recorded on a predesigned case report form in accordance with the study protocol.

Ethical Considerations:

Only patients who provide written informed consent and are willing to participate will be included.

Participants' confidentiality will be strictly maintained. Standard perioperative care will not be compromised for study purposes. All patients will be monitored for adverse events, including complications potentially related to PRP application or surgery. Any adverse events will be recorded and reported according to hospital and regulatory guidelines.

The study protocol has been submitted for approval to the Hospital Ethics Committee and the Advance Research Committee.

Study Start/Completion Dates:

Study Start Date: July 07 2022 (Actual) Primary Completion Date: January 07 2023 (Actual) Study Completion Date: February 28 2023 (Actual)

Location:

Department of cardiac surgery, PIMS.

Sponsor:

Shaheed Zulfiqar Ali Bhutto Medical University

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 to 72 years,

undergoing median sternotomy for CABG surgery.

Able and willing to provide informed consent.

Exclusion Criteria:

* Known Diabetics,

Patients unable or ineligible to donate blood for standard blood bank procedures, which includes those with low hemoglobin, blood disorders, infections, or other medical conditions preventing safe blood collection

Patients from whom autologous platelet-rich plasma (PRP) cannot be obtained due to low platelet counts, blood disorders, or other technical/medical reasons

Cardiopulmonary bypass (CPB) time > 72.5 minutes

Bilateral internal mammary artery harvested

Body Mass Index (BMI) < 18.5 or > 24.9

Active smokers

Chronic lung disease

Osteoporosis

Current steroid therapy

Ages: 45 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Superficial & Deep Sternal Wound Infections, Delayed Wound Healing and readmission. | Up to 30 days postoperatively
  Superficial Sternal Wound Infection (Defined as infection limited to skin and subcutaneous tissue within 30 postoperative days, not involving the sternum, requiring local wound care and antibiotic therapy or Vacuum Assisted Closure VAC therapy. Unit of Measure: Number of participants)
  Deep Sternal Wound Infection (Diagnosis will be made in patients developing one or more of the following within 30 postoperative days: positive culture of mediastinal tissue or fluid; clinical evidence of mediastinitis during sternal reoperation; or chest pain, sternal instability or purulent mediastinal discharge associated with a positive blood culture. Unit of Measure: Number of participants)
  Delayed Healing (Defined as failure of skin, subcutaneous tissue, or sternum to heal within 14 days after surgery. Unit of Measure: Number of participants)
  Readmission (Defined as any hospital readmission within 30 days of discharge related to the index surgery. Unit of Measure: Number of participants)

SECONDARY OUTCOMES:
Cost of hospitalization | From surgery to hospital discharge, up to 30 days postoperatively
  Total cost of care during hospital stay, including postoperative care, and medications.

OTHER OUTCOMES:
Length of ICU stay and more than 4 units of red cell count (RCC) & platelets used | Up to 30 days postoperatively
  Duration of postoperative intensive care unit (ICU) stay within 30 days following surgery. Requirement for transfusion of more than four units of red cell count (RCC) and more than four units of platelets within 30 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeen Khan Wazir, MBBS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Islamabad/Punjab, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT07352020/Prot_001.pdf